CLINICAL TRIAL: NCT04482751
Title: An Observational Single Center Study to Identify the Relationship Between Serum AMH Dynamics and Early or Normal Ovarian Response to Corifollitropin Alfa (ACO Study)
Brief Title: The Relationship Between Serum AMH Dynamics and Early or Normal Ovarian Response to Corifollitropin Alfa
Acronym: ACO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Antonio La Marca, Professor, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 184/2020
Record Dates: First submitted 2020-07-03; First posted 2020-07-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infertile women: the group consists of 80 infertile patients undergoing IVF
  Interventions: Drug: Corifollitropin alfa

INTERVENTIONS:
Drug: Corifollitropin alfa — AMH will be measured during ovarian stimulation with corifollitropin alfa
  Other Names: no other interventions

SUMMARY:
The objective of this study is to evaluate the trend of serum AMH during IVF (in vitro fertilization) cycles, in particular the possible relationship between the dynamics of AMH and the early or normal response to therapies for controlled ovarian stimulation with corifollitropin alfa. The secondary objective is to study the association between the number of follicles equal to or greater than 17 mm on the eighth day of ovarian stimulation and the decline in AMH, and to assess the predictability of the need to add additional therapies after the first week of stimulation ovarian.

DETAILED DESCRIPTION:
The study is observational and it is monocentric, and it will involve 80 patients. Patients' data, extrapolated from the medical records of the Department of Reproductive Medicine in the Policlinico Hospital in Modena, will be collected in an internal database for analysis. The inclusion criteria for the population included in the study will be: 1) basal serum FSH concentration below 20 UI/L; 2) age between 18 and 46 years; 3) body weight > 60 kg; 4) use of corifollitrofin alpha for ovarian stimulation. The following parameters will be evaluated: the age of the patients, their weight, their body mass index (BMI), duration of infertility, cycle characteristics; basal (day 2) AMH, AFC measurement, basal estradiol, basal progesterone, basal FSH, basal LH, and those same values on day 5 and day 8 of ovarian stimulation; follicles ≥ 17 mm on day 8, type of gonadothropin further added, days of stimulation with the further gonadothropin and its units per day, AMH on trigger day and the number of oocytes retrieved. The confidentiality of the informations will be guaranteed by anonymized data analysis. All the data are commonly recorded in our clinical practice.

The observed period will be of 12 months. The date of conclusion of the study, after favorable opinion of the Ethics Committee and the authorization of the Company Management, is scheduled for June 2021.

To guarantee the consent and the information of the patients involved in the study, the Information Sheet and the relative Consent Form are attached. We consider appropriate to inform the General Physician of the enlisted patients about the study: the Information Letter for the General Physician is therefore attached.

Variables/Time Points of Interest

The variables which will be recorded on cycle day 2 of a spontaneous menstruation (stimulation day 1 with Corifollitropin alfa) are: woman's age (years), weight (kg), body-mass-index (kg/m2), duration of infertility (months), cycle length (in days, by patient recall), cycle regularity (yes/no; deviation of > 5 days from two consecutive cycles is considered an irregular cycle), total number of antral follicles (2-10 mm) in both ovaries (AFC) measured by a transvaginal scan and serum AMH (ng/ml), oestradiol, progesterone, FSH and LH.

Patients will return every two days to the clinic for a transvaginal ultrasound from stimulation day 5 up to and including the day of hCG. Serum hormone concentrations (FSH, LH, oestradiol, progesterone and AMH) will be measured on stimulation days 5 and 8 and on the day of hCG.

All hormones reported above will be measured in the central lab of the ospital as per routine practice. Remaining serum will be used for the AMH assay. The measurement of the AMH will ber profrmed in the ObGyn University research Lab.

ELIGIBILITY:
Inclusion Criteria:

* basal serum FSH concentration below 20 UI/L
* age between 18 and 46 years
* body weight > 60 kg
* use of corifollitrofin alpha for ovarian stimulation.

Exclusion criteria:

* contraindications to IVF
* irregular menstrual cycles

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in serum Antimullerian Hormone (AMH) levels during ovarian stimulation | AMH will be measured at day 2, day 5, day 8 and the last day (usually day 11) of ovarian stimulation
  Serum concentrations of AMH will be measured during ovarian stimulation with corifollitropin alfa.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio La Marca, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Policlinico di Modena, Modena, Modena - MO, Italy

IPD SHARING:
Plan to Share IPD: Undecided